CLINICAL TRIAL: NCT06149871
Title: Effectiveness of Individual Physical Activity Programs to Prevent and Slow Progression of Sarcopenia and Frailty Among Thai Community-dwelling Older Adults: A Double-blind Randomized Clinical Trial
Brief Title: Effectiveness of Individual Physical Activity Programs to Prevent Sarcopenia and Frailty Among Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Thailand (Other Government)
Collaborators: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Visaratana Therakomen, Deputy Director for Academic Affairs of Bureau of Nutrition, Department of Health, Ministry of Health, Thailand
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MOHThailand
Record Dates: First submitted 2023-09-26; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Sarcopenia; Frailty
MeSH Terms: conditions — Sarcopenia; Frailty | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The Experimental groups or physical activity groups were assigned to three groups based on their muscle mass: normal, probable sarcopenia, and sarcopenia groups. The volunteers were provided with instructions on individual physical activities to be practiced at home for 30 weeks, 2-5 days per week and 50 minutes per session. These physical activities consisted of flexibility exercise for 10 minutes, aerobic exercise for 20 minutes, and resistance exercise for 20 minutes, as outlined in supplement 1. The volunteers were instructed on exercise techniques and physical activities by either sports scientists or registered nurses, and caregivers such as relatives or staff from the social club for older adults were allowed to be present during practice.
  Interventions: Behavioral: Physical activity
- Control (No Intervention): The control group did not receive any intervention apart from general suggestions and continued with their usual daily activities.

INTERVENTIONS:
Behavioral: Physical activity — resistance, aerobic, and flexibility exercises
  Arms: Intervention

SUMMARY:
Sarcopenia and frailty could be prevented and rehabilitated through individual physical activities in the form of combined exercise that could be practiced at home in daily life.

DETAILED DESCRIPTION:
The volunteers were randomly assigned to either the intervention or control group using sealed envelopes containing documents marked with either IG (intervention group) or CG (control group). The intervention group received training, after which they demonstrated and practiced the physical activities. They were provided with an exercise leaflet for self-practice at home and were followed up by phone, LINE application, and leaders of social club for older adults at least once a week to ensure regular practice. The older adults' relatives and caregivers were also trained and encouraged to practice with them in a 1:1 match. Support techniques and warning signs for stopping or taking a break during exercise were added to each posture, along with suggestions for suitable environmental management, such as flat plains, sufficient light, and no barriers within 2 meters, to reduce the risks of accidents. However, the control group did not receive any intervention apart from general suggestions and continued with their usual daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 60 and 80 years.
* Those who are able to walk independently or with the aid of walking devices.

Exclusion Criteria:

* Participants with leg or foot amputations.
* Participants who had been admitted to hospitals in the past 6 months.
* Those with underlying medical conditions such as heart disease, bone and muscle injuries, and infectious diseases.
* Individuals who did not pass the Physical Activity Readiness Questionnaire (PAR-Q).

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
The status of sarcopenia aligns with the criteria set by the Asian Working Group for Sarcopenia (AWGS). | 30 weeks
  Sarcopenia status was assessed through three aspects, including a muscle strength test using handgrip strength measured with a dynamometer, a physical performance test using the Short Physical Performance Battery (SPPB), and an appendicular skeletal muscle mass (ASM) test measured with the ACCUNIQ BC 380 tool based on bioelectrical impedance analysis (BIA). The results were aligned with the standards set by the Asian Working Group for Sarcopenia (AWGS). Sarcopenia was diagnosed by low ASM with low muscle strength or low physical performance, dynapenia was diagnosed by low muscle strength only, and pre-sarcopenia was diagnosed by low ASM or low physical performance. Participants underwent assessments both at the beginning and at the 30-week endpoint.
Muscle strength | 30 weeks
  Muscle strength, specifically handgrip strength, was measured using a hand-held dynamometer. Participants gripped the dynamometer with their dominant hand while standing, maintaining their upper arm close to the body and their elbow bent to 90 degrees, exerting maximum force. This test was conducted twice, and the superior result was recorded. Low muscle strength was diagnosed if the handgrip strength was < 26 kilograms in males and < 18 kilograms in females. Participants underwent assessments at both the beginning and the 30-week endpoint.
Physical performance | 30 weeks
  The physical performance test utilized the Short Physical Performance Battery (SPPB) to evaluate physical function, with a maximum score of 12 points. Low physical performance was diagnosed if the SPPB score was ≤ 9. Participants underwent assessments at both the beginning and the 30-week endpoint.
Muscle mass | 30 weeks
  Appendicular skeletal muscle mass (ASM) was measured using the ACCUNIQ BC 380 tool based on bioelectrical impedance analysis (BIA), and the Skeletal Muscle Mass Index (SMI) was calculated by dividing ASM in kilograms by the height in meters squared. Low muscle mass is diagnosed if SMI is < 7.0 kilograms/meter^2 in men and < 5.47 kg/m^2 in women. Participants underwent assessments at both the beginning and the 30-week endpoint.

SECONDARY OUTCOMES:
Physical frailty status based on the 5 criteria of frailty phenotype, as defined by Fried et al. 2001. | 30 weeks
  Frailty phenotype assessment followed Fried et al.'s (2001) criteria, including weakness, slowness, unintentional weight loss, exhaustion, and low physical activity. Participants were categorized as "frail" if they met three or more criteria, "pre-frail" with one or two, and "robust" if none were fulfilled.
  (i) Weakness: Handgrip strength measured with a dynamometer. (ii) Slowness: Assessed by the time taken in a 15-feet walk test. (iii) Unintentional Weight Loss: Evaluated by recording weight loss exceeding 10 pounds or 5% in the last 3 months.
  (iv) Exhaustion: Assessed with two questions from the CES-D depression scale. (v) Low Physical Activity: Determined by asking about the frequency of moderate physical activities in the past week.
  Participants underwent assessments at both the beginning and the 30-week endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Visaratana Therakomen, Diploma, Principal Investigator — Department of Health, Ministry of Public Health
Locations (1):
- Regional Health Promotion Center 2 Phitsanulok, Phitsanulok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Yes: There is a plan to make IPD and related data dictionaries available : all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Starting 6 months after publication
Access Criteria: 1. Access Criteria:
     * Ethical Approval: Requestors must provide evidence of ethical approval from their respective institutions or review boards for the proposed analyses.
     * Data Security Measures: Researchers must demonstrate the implementation of robust data security measures to protect the confidentiality and integrity of the shared data.
  2. Additional Supporting Information:
     * Study Protocol: A detailed study protocol outlining the objectives, methodologies, and analysis plan must be submitted along with the request for IPD access.
     * Data Dictionary: A comprehensive data dictionary defining variables, codes, and any transformations applied to the data should accompany the request.
URL: https://nutrition2.anamai.moph.go.th/th/research2

REFERENCES:
- [Background] Cadore EL, Casas-Herrero A, Zambom-Ferraresi F, Idoate F, Millor N, Gomez M, Rodriguez-Manas L, Izquierdo M. Multicomponent exercises including muscle power training enhance muscle mass, power output, and functional outcomes in institutionalized frail nonagenarians. Age (Dordr). 2014 Apr;36(2):773-85. doi: 10.1007/s11357-013-9586-z. Epub 2013 Sep 13. PMID 24030238
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Dent E, Morley JE, Cruz-Jentoft AJ, Arai H, Kritchevsky SB, Guralnik J, Bauer JM, Pahor M, Clark BC, Cesari M, Ruiz J, Sieber CC, Aubertin-Leheudre M, Waters DL, Visvanathan R, Landi F, Villareal DT, Fielding R, Won CW, Theou O, Martin FC, Dong B, Woo J, Flicker L, Ferrucci L, Merchant RA, Cao L, Cederholm T, Ribeiro SML, Rodriguez-Manas L, Anker SD, Lundy J, Gutierrez Robledo LM, Bautmans I, Aprahamian I, Schols JMGA, Izquierdo M, Vellas B. International Clinical Practice Guidelines for Sarcopenia (ICFSR): Screening, Diagnosis and Management. J Nutr Health Aging. 2018;22(10):1148-1161. doi: 10.1007/s12603-018-1139-9. PMID 30498820
- [Background] Dent E, Morley JE, Cruz-Jentoft AJ, Woodhouse L, Rodriguez-Manas L, Fried LP, Woo J, Aprahamian I, Sanford A, Lundy J, Landi F, Beilby J, Martin FC, Bauer JM, Ferrucci L, Merchant RA, Dong B, Arai H, Hoogendijk EO, Won CW, Abbatecola A, Cederholm T, Strandberg T, Gutierrez Robledo LM, Flicker L, Bhasin S, Aubertin-Leheudre M, Bischoff-Ferrari HA, Guralnik JM, Muscedere J, Pahor M, Ruiz J, Negm AM, Reginster JY, Waters DL, Vellas B. Physical Frailty: ICFSR International Clinical Practice Guidelines for Identification and Management. J Nutr Health Aging. 2019;23(9):771-787. doi: 10.1007/s12603-019-1273-z. PMID 31641726
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Result] Afilalo J. Conceptual Models of Frailty: The Sarcopenia Phenotype. Can J Cardiol. 2016 Sep;32(9):1051-5. doi: 10.1016/j.cjca.2016.05.017. Epub 2016 Jun 2. PMID 27568870